CLINICAL TRIAL: NCT06654349
Title: Short-term Recovery After Trapeziectomy and TMC Prosthesis: a Diary Study
Acronym: THUMB Diary
Status: Recruiting | Type: Observational
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: OC-2024-001; N24.085 (Other: METC LDD)
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Arthrosis of First Carpometacarpal Joint
Keywords: Trapeziectomy; Diary; TMC-arthroplasty; Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Trapeziectomy: This cohort consist of patients receiving a trapeziectomy for arthrosis of the first carpometacarpal joint. The cohort will include 100 patients
- TMC-arthroplasty: This cohort consist of patients receiving TMC-arthroplasty for arthrosis of the first carpometacarpal joint. The cohort will include 100 patients

SUMMARY:
Rationale: The trapeziometacarpal (TMC) joint is one of the most common areas in the hand and wrist to develop osteoarthritis (OA). Currently, the two most widely used procedures are the trapeziectomy and the TMC-joint arthroplasty, both with their own pros and cons. No studies have demonstrated superiority of TMC-joint arthroplasty over gold-standard trapeziectomy. And no clinical studies show short-term recovery and patient experience after trapeziectomy or TMC-joint arthroplasty.

Objective: To gather insight in short-term recovery and patient experience after a trapeziectomy or TMC prosthesis regarding pain, pain medication, function and quality of life.

Study design: A prospective observational cohort diary study.

Study population: In total 200 subjects with TMC-joint osteoarthritis will participate: 100 subjects will have trapeziectomy and 100 subjects will have TMC-joint arthroplasty

Main study parameters/endpoints: The main study parameters are the pain, function and quality of life during the first 8 weeks after surgery.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will have no direct benefit from participation in this study. Subjects will only complete a diary and questionnaires for this study. Therefore, we expect no risks from participation. The burden for subjects consists of approximately five minutes daily for the diary in the first eight weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Failed conservative treatment for osteoarthritis
* Planned for trapeziectomy or TMC-joint arthroplasty
* Age 18-75 years
* Willing and able to comply with the postoperative functional assessment and to participate in a rehabilitation schedule

Exclusion Criteria:

* Mentally disabled patients
* Active infection
* Current malignancy
* Infiltration (corticoids < 3 months)

The following criteria is specific for the TMC-joint arthroplasty group and is an addition to the criteria mentioned above:

* Trapezium height < 8 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive eligible subjects will be asked to participate and devided into either the Trapeziectomy cohort or the TMC-arthroplasty cohort, depending on the scheduled operative treatment for the osteoarthrosis of the first carpometacarpal joint.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain | 8 weeks
  Pain will be measured each day in a diary for the first 8 weeks after surgery with the Numeric Rating Scale for Pain (NRS), which is a scale ranging from zero to ten on which patients can score their pain. It is a widely used instrument in varying populations due to its ease of administration and clinical relevance to the subject.
Function | 8 weeks
  Function will be measured each week in a diary for the first 8 weeks after surgery with the The Patient-Related Wrist/Hand Evaluation (PRWHE), which is a 15-item questionnaire concerning pain and function. Subjects are able to rate their pain and disabilities from zero to ten.
Quality of life (QoL) | 8 weeks
  QoL will be measured twice a week in a diary for the first 8 weeks after surgery with the EQ-5D, which is a general health-related quality-of-life questionnaire and consists of five questions regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression and one visual analog scale (VAS) to document the perceived quality of life. It is also used to assess quality of life adjusted life years (QALY).

SECONDARY OUTCOMES:
Complications | 1 year
  Complications will be measured in the number of complications.
Pain medication | 8 weeks
  Pain medication will be measured with a diary during the first 8 weeks after surgery
PROMs - NRS | 1 year
  Patient-related outcome measurements (PROMs) will be measured with the NRS as part of the standard care. Numeric Rating Scale for Pain (NRS) is a scale ranging from zero to ten on which patients can score their pain. It is a widely used instrument in varying populations due to its ease of administration and clinical relevance to the subject.
PROMs - PRWHE | 1 year
  Patient-related outcome measurements (PROMs) will be measured with the PRWHE as part of the standard care. The Patient-Related Wrist/Hand Evaluation (PRWHE) is a 15-item questionnaire concerning pain and function. Subjects are able to rate their pain and disabilities from zero to ten.
PROMs - EQ5D | 1 year
  Patient-related outcome measurements (PROMs) will be measured with the EQ5D as part of the standard care. EQ-5D is a general health-related quality-of-life questionnaire and consists of five questions regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression and one visual analog scale (VAS) to document the perceived quality of life. It is also used to assess quality of life adjusted life years (QALY). It has been translated into Dutch and validated in different populations.
PROMs - HADS | 1 year
  Patient-related outcome measurements (PROMs) will be measured with the HADS as part of the standard care. The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire concerning the mental state of the subject (i.e. anxiety and depression).

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided